CLINICAL TRIAL: NCT04860635
Title: An Open Label Safety Study of a Single Administration of F14 in Patients Undergoing Unilateral Total Knee Replacement
Brief Title: Safety of F14 Following Total Knee Replacement
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study superseded by alternative Phase 3 trial
Sponsor: Arthritis Innovation Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100-CIP03-P
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-02

CONDITIONS: Analgesia
Keywords: total knee arthroplasty; postoperative pain; NSAID; multimodal analgesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- F14 (sustained release celecoxib) (Experimental): Intra-articular F14 administration immediately following TKR surgery, and concurrent with multimodal standard of care analgesia
  Interventions: Drug: F14 (sustained release celecoxib)

INTERVENTIONS:
Drug: F14 (sustained release celecoxib) — Celecoxib in BEPO® drug delivery system

SUMMARY:
Open-label single-arm study in which all subjects receive F14 as part of a scheduled TKR and multimodal analgesia

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or females indicated for primary, unilateral TKR
2. Between 45-80 years of age
3. Capable of giving signed informed consent
4. Body Mass Index (BMI) ≤ 40 kg/m2
5. Medically stable as determined by the Investigator, based on physical examination, clinical laboratory tests, and 12-lead ECG findings, as well as medical history from subject and pre-study source documents from other care providers
6. Absence of fixed flexion deformity exceeding 15deg
7. Absence of varus or valgus deformity exceeding 15deg
8. Minimum pre-operative flexion arc of 100deg
9. American Society of Anesthesiologists Physical Status Classification System (ASA-PSC) score ≤ 3
10. Females of childbearing potential with a negative serum pregnancy test at screening or males with a partner that is of childbearing potential, who agree to employ adequate birth control measures for the full duration of the study
11. Has undergone successful total knee replacement surgery, which in the opinion of the Investigator, will not affect the subject's study follow-up

Exclusion Criteria:

1. Known allergy or hypersensitivity to active ingredient celecoxib, OR known allergy or hypersensitivity to sulfonamide antibiotics or sulfa containing drugs when an allergy to celecoxib is unknown
2. Unwilling or unable to discontinue use of nonsteroidal anti-inflammatory drugs (NSAIDs) within 7 days of scheduled surgery, or medical marijuana or cannabidiol (CBD) within 10 days
3. Total or partial knee arthroplasty in the contralateral knee < 6 months prior to study surgery
4. Participation or scheduled participation in another clinical study involving an investigational drug or device within 30 days before screening or during study follow-up
5. Active or past infection in the index knee
6. Documented osteonecrosis of the index knee within previous 12 months
7. Other planned major surgery within 12 months of study surgery
8. Had a malignancy in the last year, except for non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
9. Diagnosis of skin disorders including psoriasis, vascular insufficiency ulcers, and chronic venous stasis
10. History of coronary or vascular stent placed within 3 months
11. Suspected opioid abuse in the last 12 months with a score exceeding 5 on the DAST-10 questionnaire, and/or taking opioids on most days in the past three months, and currently taking >120 mg morphine equivalent dose (MED) at least 5 days per week in the month prior to screening
12. Current medical diagnosis or subject-reported seizure disorder
13. Current peripheral neuropathy
14. History of complex regional pain syndrome (CRPS)
15. Diagnosis of clinically significant liver hepatic and/or renal abnormalities within previous 2 years
16. Diagnosis of diabetes with HbA1c ≥7%
17. Current inflammatory arthritides (e.g., rheumatoid arthritis, lupus erythematosus, ankylosing spondylitis, psoriatic arthritis), or traumatic bone injuries within 12 months before scheduled surgery, except for clinically stable/non-active gout that does not affect the knee and does not interfere with walking
18. Treatment with immunosuppressants, antipsychotics, anticholinergics, or anticonvulsants within 1 month of intervention (antipsychotic stable dosage established for >30 days will be allowed)
19. Current or historical evidence of any clinically significant disease or condition, especially cardiovascular, pulmonary, or neurological
20. Participation in active or pending personal injury or workers' compensation litigation

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | From Day 0 to 12 months

OTHER OUTCOMES:
NRS pain intensity | From Day 1 to 3 months
  Numerical rating scale (NRS); 11-point scale ranges from '0' representing "no pain" to '10' representing "worst imaginable pain"
Duration of need for walking aids | From Day 1 to 3 months
Proportion of subjects using concomitant analgesics at any timepoint | From Day 1 to 3 months
Celecoxib concentration in plasma | At specified timepoints up to 3 months
  PK sub-study in 15 participants

CONTACTS AND LOCATIONS:
Overall Officials: Jared Foran, MD, Principal Investigator — Panorama Orthopedics & Spine Center
Locations (2):
- United States (2):
  - Panorama Orthopedics & Spine Center, Denver, Colorado
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No